CLINICAL TRIAL: NCT05532618
Title: Efficacy of Adductor Canal Block for Anterior Cruciate Ligament Surgery: A Prospective Double Blinded Randomized Controlled Trial
Brief Title: Efficacy of Adductor Canal Block for Anterior Cruciate Ligament Surgery
Acronym: DUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Leon Timmerman, M.D., PhD, principal investigator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NL 81489.100.22
Record Dates: First submitted 2022-09-02; First posted 2022-09-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: adductor canal block
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Levobupivacaine

STUDY DESIGN:
Intervention Model Description: Patients are randomized to receive an intervention (nerve block) with either an active drug or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Medication is prepared by study personell not otherwise involved in the study according to a computer generated randomization plan. This plan will be available for analyses after the study. Primary investigator is able to retreive the allocation prematurely if indicated (emergency).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levobupivacaine (Active Comparator): Intervention group; 10 ml of Levobupivacaine 0.25% will be added in the adductor canal using ultrasound
  Interventions: Procedure: Adductor canal block; Drug: Levobupivacaine
- Placebo (Placebo Comparator): Control group; 10 ml of sodium chloride 0.9% will be added in the adductor canal using ultrasound
  Interventions: Procedure: Adductor canal block; Drug: Placebo

INTERVENTIONS:
Procedure: Adductor canal block — Before anterior cruciate ligament surgery an adductor canal block will be placed using ultrasound.
Drug: Levobupivacaine — Levobupivacaine
  Arms: Levobupivacaine
Drug: Placebo — 10 ml of sodium chloride 0.9%
  Arms: Placebo

SUMMARY:
The goal of this study is to objectify the postoperative pain level, the use of opiates and postoperative nausea and vomiting after adding the adductor canal block to the standard pain regiment after anterior cruciate ligament surgery

DETAILED DESCRIPTION:
Patients scheduled for anterior cruciate ligament surgery will be randomized in an intervention and control group following informed consent.

Before surgery, patients will receive an adductor canal bock with Levobupivacaine (intervention group) or 0.9% saline (control group).

Following surgery, pain intensity, analgesic consumption and pain satisfaction will be recorded bij patients in a diary for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Undergoing anterior cruciate ligament surgery under general anesthesia
* ASA I-III

Exclusion Criteria:

* Contraindication for locoregional anesthesia; infection at the target puncture site, allergy to local anesthetics,
* Neuromuscular disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain level | Within first 48 hours after surgery
  Using Numerical Rating Scales for pain from 1 to 10, 1 is no pain, 10 is the worst pain you can imagine

SECONDARY OUTCOMES:
Opiate use | Within first 48 hours after surgery
  postoperative use of opiates (Morphine equivalent dose (mg))
Nausea | Within first 48 hours after surgery
  Postoperative nausea (yes/no)
Block result | within first 24 hours after surgery
  If there's any loss of motor function (no quadriceps paresis, partial quadriceps paresis, complete quadriceps paresis.) using bromage score
Patient satisfaction | 48 hours after surgery
  Using Numerical Rating Scales from 1 to 10, 1 is not satisfied at all, 10 is completely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Leon Timmerman, dr, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Following publication of the results, anonymized IPD (all study results) will be available for meta-analyses upon request.
Supporting Information: Study Protocol
Time Frame: Following publication of the results, for at least 15 years.
Access Criteria: Data will be available on request. If a journal allows online sharing of IPD with a publication, this will be considered as well.

REFERENCES:
- [Background] Kwofie MK, Shastri UD, Gadsden JC, Sinha SK, Abrams JH, Xu D, Salviz EA. The effects of ultrasound-guided adductor canal block versus femoral nerve block on quadriceps strength and fall risk: a blinded, randomized trial of volunteers. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):321-5. doi: 10.1097/AAP.0b013e318295df80. PMID 23788068
- [Background] Johnston DF, Sondekoppam RV, Uppal V, Litchfield R, Giffin R, Ganapathy S. Effect of combining peri-hamstring injection or anterior obturator nerve block on the analgesic efficacy of adductor canal block for anterior cruciate ligament reconstruction: a randomised controlled trial. Br J Anaesth. 2020 Mar;124(3):299-307. doi: 10.1016/j.bja.2019.11.032. Epub 2020 Jan 21. PMID 31980156